CLINICAL TRIAL: NCT02122744
Title: Randomised Placebo Controlled Trial of rTMS Quadri Pulse Over Visual Cortex for the Prevention of Chronic Migraine
Brief Title: RCT Versus Placebo of rTMSQP Over Visual Cortex for the Prevention of Chronic Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Full Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CB-1331
Record Dates: First submitted 2013-11-04; First posted 2014-04-25 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Super Rapid Magstim Stimulator rTMS QP (Active Comparator): rTMS QP is delivered over the visual cortex for 30 minutes, 2 times a week for 8 weeks, in 15 patients
  Interventions: Device: Super Rapid Magstim Stimulator
- Placebo (Placebo Comparator): rTMS QP placebo (coil perpendicular to the scalp) is delivered over the visual cortex for 30 minutes, 2 times a week for 8 weeks, in 15 patients.
  Interventions: Device: Super Rapid Magstim Stimulator (sham)

INTERVENTIONS:
Device: Super Rapid Magstim Stimulator — The repetitive transcranial magnetic stimulation (rTMS) is able to modify cortical excitability and reactivity. 1Hz rTMS inhibits the cortex, 10Hz excites it. In particular, a new paradigm of rTMS, the rTMS quadri pulse has a more lasting and effective activity.
  The side effects are rare and transient: migraine,contractions of the muscles of the neck due to muscle stimulation by the electromagnetic field of the coil.
  Arms: Super Rapid Magstim Stimulator rTMS QP
Device: Super Rapid Magstim Stimulator (sham) — coil perpendicular to the scalp
  Arms: Placebo

SUMMARY:
Evaluation of inhibiting rTMS QP over the visual cortex for the prevention of chronic migraine. The aim of the study is to confirm that inhibiting rTMS QP is capable to decrease the frequency of migraine and if its effect is stronger than placebo effect.

DETAILED DESCRIPTION:
The investigators have already inquired if inhibiting rTMS QP over the visual cortex determines a reduction of frequency of migraine in a previous study. After 2 weekly sessions for a month, the investigators demonstrated a reduction of 47% in migraine frequency. In this study, the investigators aim to compare rTMS QP effect with the placebo effect and to evaluate if rTMS QP is capable to induce changes in VEP, CHEPS and QST.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic migraine (ICHD III beta 1.3) with or without medication overuse.

Exclusion Criteria:

* other diseases or contraindication for the magnetic stimulation (epilepsy, pacemaker, metallic prothesis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Frequency of migraine | 12 months
  The investigators evaluate the frequency of migraine during the treatment and 2 months after its end.

SECONDARY OUTCOMES:
Intensity of migraine | 12 months
  The investigators evaluate the intensity of migraine during the treatment and 2 months after its end
Acute medication intake | 12 months
  The investigators evaluate acute medication intake during the treatment and 2 months after its end
Attack duration | 12 months
  The investigators evaluate attack duration during the treatment and 2 months after its end
Scores on psychological scales | 12 months
  The investigators evaluate scores on psychological scales during the treatment and 2 months after its end

CONTACTS AND LOCATIONS:
Overall Officials: Jean Schoenen, HP, Principal Investigator — University of Liege; Delphine Magis, MD,PhD, Principal Investigator — University of Liege
Locations (1):
- Roberta Baschi, Liège, Belgium